CLINICAL TRIAL: NCT04404075
Title: Skin Tracker: A Mobile Health App to Monitor Skin Disease Activity and Treatment Use
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 19-28676
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 patients: 1. Age 18 and above
  2. Eczema Area and Severity Index (EASI) score ≥ 10
  3. Investigator Global Assessment (IGA) ≥ 3
  Interventions: Other: SkinTracker Mobile App
- Group 2 patients: 1. Age 18 and above
  2. Eczema Area and Severity Index (EASI) score ≥ 1 but < 10
  3. Investigator Global Assessment (IGA) 1 or 2
  Interventions: Other: SkinTracker Mobile App
- Group 3 patients: 1. Age 12 to 17
  2. Eczema Area and Severity Index (EASI) score ≥ 10
  3. Investigator Global Assessment (IGA) ≥ 3
  Interventions: Other: SkinTracker Mobile App
- Group 4 patients: 1. Age 12 to 17
  2. Eczema Area and Severity Index (EASI) score ≥ 1 but < 10
  3. Investigator Global Assessment (IGA) 1 or 2
  Interventions: Other: SkinTracker Mobile App

INTERVENTIONS:
Other: SkinTracker Mobile App — a research-oriented eczema app to longitudinally track atopic dermatitis severity, symptoms, quality of life, physical activity, medication usage, and adverse events in a real-world setting

SUMMARY:
Design and beta-test a research-oriented mobile health app to assess disease activity, quality of life, treatment patterns, adverse medication effects, and lifestyle factors in patients with atopic dermatitis.

DETAILED DESCRIPTION:
Mobile health technology, including smartphone apps and wearable monitors, has tremendous potential to transform clinical research. Recording of patient outcomes on a smartphone device and camera in the home setting can greatly reduce the number of in person research visits, saving tremendous costs, time, and effort associated with data entry. This also allows for easier recruitment of study subjects, who can be enrolled in geographic locations beyond academic research centers. After FDA approval of a therapy, mobile health technology can help researchers understand how that particular therapy is being used in a real-world setting, including frequency of use, adverse events, and impact of use on disease symptoms and patient quality of life. In this study, the investigators will create a mobile app to help the atopic dermatitis community understand the types of data and quality of data that can be gathered from atopic dermatitis patients longitudinally. A review of existing atopic dermatitis mobile apps on the market reveals they are consumer-oriented and may not be able to fully capture high-quality research data. The investigator proposed app is specifically geared for research, and thus fills an important gap. The research team will develop SkinTracker, a research-oriented eczema app to longitudinally track atopic dermatitis severity, symptoms, quality of life, physical activity, medication usage, and adverse events in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and comply with the protocol.
2. At least 13 years of age.
3. Diagnosis of atopic dermatitis by dermatologist for at least 6 months.
4. Physical exam within clinically acceptable limits.
5. Own or have access to a mobile device that is compatible with study mobile application SkinTracker.

Exclusion Criteria:

1. Subject is unable to provide written informed consent or comply with the protocol.
2. Unable to input data into SkinTracker mobile app.
3. Subject is younger than 13 years of age.
4. Serious known infection.
5. History of immunosuppression (including human immunodeficiency virus (HIV)).
6. History of malignancy within 5 years prior to screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
7. Severe concomitant illness.
8. Physical exam not within clinically acceptable limits.
9. Subjects possess other diagnoses that, in the investigator's opinion, preclude him/her from safely participating in this study or interfere

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-center, observational, pilot study. Ten subjects with atopic dermatitis will be enrolled.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Average change in eczema area and severity index EASI score at month 6 | Month 6
  Patient eczema area and severity index (EASI) will be measured. It is a tool for measuring the amount and severity of eczema a patient has on his or her body, scale is 0-72, 0 means clear and 72 means severe eczema

SECONDARY OUTCOMES:
Average change in eczema area and severity index EASI score at month 3 | Month 3
  Patient eczema area and severity index (EASI) will be measured. It is a tool for measuring the amount and severity of eczema a patient has on his or her body, scale is 0-72, 0 means clear and 72 means severe eczema
Average change in Investigator global assessment (IGA) at month 6 | Month 6
  Patient Investigator global assessment (IGA) score will be measured from 12 to 18 months, it is a scale to estimate overall severity of eczema but does not take into account BSA specifically, scale is 0 to 4, 0 is clear and 4 is severe
Average change in Investigator global assessment (IGA) at month 3 | Month 3
  Patient Investigator global assessment (IGA) score will be measured from 12 to 18 months, it is a scale to estimate overall severity of eczema but does not take into account BSA specifically, scale is 0 to 4, 0 is clear and 4 is severe

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No